CLINICAL TRIAL: NCT03115762
Title: Pharmacokinetics,Safety and Immunogenicity of ASKB1202 in Chinese Healthy Subjects: a Randomized, Double-blinded, Single-dose, Parallel-arm, Active-comparator Clinical Phase I Study
Brief Title: Pharmacokinetics and Safety Study of ASKB1202 in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASK-LC-B1202-1
Record Dates: First submitted 2017-04-12; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: ASKB1202
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASKB1202 (Experimental): Subject to receive one intravenous (i.v.) infusion of ASKB1202
  Interventions: Biological: ASKB1202
- bevacizumab A (Active Comparator): Subject to receive one intravenous (i.v.) infusion of bevacizumab sold in China
  Interventions: Biological: bevacizumab
- bevacizumab B (Active Comparator): Subject to receive one intravenous (i.v.) infusion of bevacizumab sold in Europe
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — recombinant humanized monoclonal antibody produced by DNA technology in Chinese Hamster Ovary cells
  Arms: bevacizumab A; bevacizumab B
Biological: ASKB1202
  Arms: ASKB1202

SUMMARY:
This trial will investigate the pharmacokinetic,immunogenicity and safety biosimilarity of ASKB1202 compared to bevacizumab sold in China and Europe.

ELIGIBILITY:
Inclusion Criteria:

* 1.Healthy males,aged 18 to 50 years. 2.A complete medical history, including disease history,physical examination, vital signs, 12-lead electrocardiogram (ECG), and chest X-ray image.

  3.Clinical laboratory tests is normal or the abnormality is not clinical significant determined by researchers.

  4.The subjects were willing to take effective contraceptive measures within 2 months before use of the drug and 6 months after.

  5.The subjects could understand the procedures and methods of this study, were willing to strictly abide the clinical trial plan to complete the test, sign the Informed Notice.

Exclusion Criteria:

* 1.Any evidence of a historical or existing clinically relevant concomitant disease, as determined by researchers.

  2.Acute,chronic active infections during screening of the study and admission(1 day before treatment),or has a history of active tuberculosis.

  3.Hemorrhaged or donated blood (including the components of blood donation)， or received blood transfusion ≥400 mL within 3 months before screening；Hemorrhaged or donated blood (including the components of blood donation) ≥200 mL within a month before the screening .

  4.Any finding of abnormality which has clinical significance during the screening of the clinical tests determined by researchers.

  5.Currently suffering from hypertension,abnormal blood pressure during study screening and hospital admission(1 day before use of drug):systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg.

  6.Any disease causes it to increase the risk of bleeding or thrombosis, such as bleeding or thrombosis genetic predisposition, or has a history of traumatic hemorrhage, thromboembolic events, blood coagulation disease and thrombocytopenia (platelet count <100000/L) or international standardization ratio (INR) is higher than 1.44.

  7.Suffered or suffering from clinical significant atopic allergy, hypersensitivity or allergic reaction, including known or suspected sensitive to one component in drug; abnormal serum immunoglobulin E (IgE) determined by researchers.

  8.Abnormal electrocardiogram (ECG) with clinical significance, such as QTc interphase is greater than 450 milliseconds.

  9.A history of gastrointestinal perforation or any fistula. 10.Has a wound without healing or fracture in study screening and admission. 11.Orthostatic hypotension, syncope and dizziness or has a history of shock caused by any reason.

  12.Suffered from malignant tumors (except that controlled basal cell carcinoma and squamous cell carcinoma).

  13.Has been vaccinated within 4 weeks before screening , or plan to get the vaccine during the study period.

  14.Has a history of taking beacizumab or anti VEGF targeted agents or having the antibody of anti VEGF.

  15.Participated in another trial within three months prior to administration or had a monoclonal antibody therapy within twelve months prior to administration.

  16.Received a surgery within 28 days prior to administration, including dental suture or wound dehiscence, or plan to undergo surgery including dental surgery during the study and 60 days after the last administration of the protocol specified treatment.

  17.Used any drug that is harmful to major organs within 3 months before administration,or use any drug within 14 days prior to participation.

  18.Smoker who smoked >5 cigarettes per day within 3 months prior to the research and unable to refrain from smoking during the research.

  19.History of alcohol abuse(drink alcohol more than 14 units a week [1 unit = 285 mL beer or 25 mL of liquor or 100 mL of wine); positive result for alcohol breath test within 24h before treatment;or unable to refrain from drinking during the study.

  20.History of taking drugs or drug abuse;or positived result for drug screening;or unable to refrain from drug abuse during the study.

  21.Positive hepatitis b surface antigen , hepatitis c antibody , HIV antibody and syphilis antibody.

  22.Any condition that not suitable to anticipate the research or bring obvious risks to the subjects according to researchers.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 100 days
  Maximum measured concentration of the analyte in plasma
AUC0-t | up to 100 days
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point
AUC0-∞ | up to 100 days
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity

SECONDARY OUTCOMES:
Tmax | up to 100 days
  Time to peak
t1/2 | up to 100 days
  Terminal-phase elimination half-life

IPD SHARING:
Plan to Share IPD: Undecided